CLINICAL TRIAL: NCT00004443
Title: Study of NTBC for Tyrosinemia I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: 199/13443; UWASH-FDR001445
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-04

CONDITIONS: Tyrosinemia I
Keywords: inborn errors of metabolism; rare disease; tyrosinemia I
MeSH Terms: conditions — Metabolism, Inborn Errors; Rare Diseases

INTERVENTIONS:
Drug: NTBC

SUMMARY:
OBJECTIVES: I. Assess the safety and efficacy of NTBC in children with tyrosinemia I.

II. Evaluate the effects of NTBC on survival, rate of neurologic crises, improvement in renal tubular damage, reduction in the need for liver transplantation, and reduction in the development of hepatocarcinoma in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients are stratified according to age at onset of symptoms (0-2 months vs 2-6 months vs greater than 6 months).

Patients receive oral NTBC twice a day. Treatment continues in the absence of unacceptable toxicity.

Patients are followed once a month for 6 months, then every 3 months thereafter.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
* Confirmed diagnosis of tyrosinemia Detected through newborn screening before the onset of symptoms OR Diagnosed on the basis of symptoms (liver disease, neurological crises, growth failure) and succinylacetone in urine or blood and/or fumarylacetoacetate dehydratase deficiency in cultured fibroblasts or liver biopsy

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 1998-10; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: C. Ronald Scott, Study Chair — University of Washington
Locations (3):
- United States (2):
  - Oregon Health Sciences University, Portland, Oregon
  - University of Washington School of Medicine, Seattle, Washington
- Hopital Sainte Justine, Montreal, Quebec, Canada